CLINICAL TRIAL: NCT01535157
Title: Phase I/II Trial of Fenretinide/LXS Oral Powder (NSC 374551) Plus Ketoconazole in Recurrent Ovarian Cancer and Primary Peritoneal Carcinoma
Brief Title: Fenretinide/LXS Oral Powder Plus Ketoconazole in Recurrent Ovarian Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: drug combination not providing any efficacy. Will use this data in opening new trial
Sponsor: South Plains Oncology Consortium (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPOC-2011-001; NCT01550692 (obsolete NCT alias)
Record Dates: First submitted 2012-02-03; First posted 2012-02-17 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Ovarian Cancer; Cancer of Ovary; Cancer of the Ovary; Ovary Neoplasms; Primary Peritoneal Carcinoma
Keywords: Chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Ketoconazole; Fenretinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fenretinide/LXS + Ketoconozale (Experimental): One course is defined as 7 days of Fenretinide/LXS + Ketoconazole followed by 14 days of rest. A course is repeated every 21 days if no evidence of disease progression for six courses.
  Interventions: Drug: Fenretinide/LXS + Ketoconazole

INTERVENTIONS:
Drug: Fenretinide/LXS + Ketoconazole — Starting dose is: Fenretinide/LXS 800 mg 4-HPR/m2/day and Ketoconazole 400 mg/day
  Other Names: 4-HPR; N-(4-hydroxyphenyl)retinamide; Nizoral; Feoris

SUMMARY:
The purpose of this study is to determine the effectiveness of fenretinide (4-HPR/LXS) plus ketoconazole in the treatment of recurrent ovarian cancer or primary peritoneal carcinoma. In addition, researchers would like to determine if the drugs are most effective together or if fenretinide (4-HPR/LXS) is most effective alone.

DETAILED DESCRIPTION:
In this study, an initial Phase I component of six patients will be conducted to monitor for potential toxicities as this wil be the initial adult experience of fenretinide (4-HPR) given together with ketoconazole

ELIGIBILITY:
Inclusion Criteria:

* Recurrent epithelial ovarian cancer or primary peritoneal carcinoma that can be platinum sensitive or platinum resistant
* SWOG Performance Status 0-2
* Previously received a platinum and paclitaxel containing regimen
* Projected Life Expectancy of at least 3 months
* Adequate bone marrow function
* Adequate organ function
* Must have received at least 1 prior salvage regimen for recurrent ovarian cancer
* Recovery from acute toxicities from surgery, radiation or chemotherapy
* At least 3 weeks from last therapy

Exclusion Criteria:

* Prior fenretinide oral capsule use allowed. If prior IV fenretinide use, must contact study chair for eligibility
* Second malignancy within last 5 years
* Use of concomitant antioxidants, such as vitamin C or E
* Untreated or symptomatic brain metastases
* History of hypertriglyceride levels > 200 mg/dl; triglyceride levels < 200 and receiving treatment are okay.
* Use of certain medications is prohibited - contact study coordinator for information

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Phase 2: Progression Free Survival | From date of enrollment until date of documented progression or date of death (up to 48 months after last patient enters treatment)
  The objective response rate will be calculated as the percent of evaluable patients whose best response is a CR or PR, and assoicated exact 95% confidence intervals will be calculated. Time to treatment failure, duration of response and survival will be estimated using the product-limit method of Kaplan and Meier.
Phase 2: Overall Survival | From enrollment up to first date of progressive disease or death from any cause (up to 48 months after last patient entered treatment)
  The objective response rate will be calculated as the percent of evaluable patients whose best response is a CR or PR, and assoicated exact 95% confidence intervals will be calculated. Time to treatment failure, duration of response and survival will be estimated using the product-limit method of Kaplan and Meier.
Phase 1: To determine the systemic toxicity profile of 4-HPR/LXS oral powder + ketoconazole | From time of first dose to the last (average 6 months)
  Toxicity information recorded will include the type, severity, time of onset, time of resolution, and the probable association with the study regimen.
Phase 2: Event Free Survival | From enrollment up to the first date of progressive disease or death from any cause (up to 48 months after last patient entered on treatment)
  The objective response rate will be calculated as the percent of evaluable patients whose best response is a CR or PR, and assoicated exact 95% confidence intervals will be calculated. Time to treatment failure, duration of response and survival will be estimated using the product-limit method of Kaplan and Meier.

SECONDARY OUTCOMES:
Pharmacokinetics - | up to 48 months after the last subject enrolled
  Area under the plasma concentration versus time curve (AUC) steady state plasma concentrations; drug levels in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Jayanthi Lea, MD, Study Chair — University of Texas Southwestern Medical Center; Barry J Maurer, MD, PhD, Study Director — Texas Tech University Health Sciences Center
Locations (3):
- United States (3):
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Click here for more information about the South Plains Oncology Consortium — http://www.sponc.org